CLINICAL TRIAL: NCT01083680
Title: Post-marketing Observational Study to Evaluate the Safety and Efficacy of HUMIRA® (Adalimumab SC) for the Treatment of Moderate to Severe Crohn's Disease in Daily Clinical Practice
Brief Title: Effectiveness and Safety in Patients With Crohn´s Disease in Clinical Routine
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-278
Record Dates: First submitted 2010-02-26; First posted 2010-03-10 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Crohn's Disease
Keywords: Routine clinical setting; Long-term efficacy and safety; Crohn's Disease; Humira®; Adalimumab
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Crohn's Disease (CD): Participants with Crohn's Disease treated with adalimumab (HUMIRA®) in routine clinical practice.

SUMMARY:
The purpose of this study was intended to evaluate the long-term safety and effectiveness of adalimumab in participants with Crohn's disease (CD) who are treated as recommended in the product label.

DETAILED DESCRIPTION:
This study was a 60-month prospective, multicenter, observational study of adalimumab in adult participants with CD who resided in Germany. Visits were scheduled every 3 months for the first year and every 6 months thereafter. Participants continued in the study for a maximum of 60 months or until discontinuation from adalimumab therapy.

ELIGIBILITY:
Inclusion Criteria:

- Severe, active Crohn's Disease in patients with insufficient response to a complete and adequate therapy of glucocorticoid and/or immunosuppressive drug and/or hypersensitivity against such a therapy or in patients where such a therapy is contraindicated.

Exclusion Criteria:

- Hypersensitivity against the drug or one of the other ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consisted of participants with Crohn's Disease (CD) who were treated with adalimumab.
Sampling Method: Non-Probability Sample
Enrollment: 4107 (Actual)
Dates: Start 2007-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Bloch, MD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4107 participants were enrolled: 1621 in the full analysis set (FAS) population were analyzed for efficacy; 4107 were analyzed for safety.
Groups:
- Participants With Crohn's Disease (CD): Participants with Crohn's Disease treated with adalimumab in routine clinical practice.
Period: Overall Study
Arm/Group | Participants With Crohn's Disease (CD)
Started | 4107
Full Analysis Set (FAS), Efficacy | 1621
Completed | 263
Not Completed | 3844
Not completed — Lost to Follow-up | 2758
Not completed — Withdrawal by Subject | 1086

BASELINE CHARACTERISTICS:
Population: Baseline analyses accounts for safety analysis set population (all participants who received at least 1 dose of study drug).
Arm/Group | Participants With Crohn's Disease (CD)
Number analyzed (Participants) | 4107
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline analysis (age, continuous) accounts for safety analysis set population with available data. This information wasn't available for 31 participants.
  years
    number analyzed (Participants) | 4076
    (all) | 36.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline analysis (gender) accounts for safety analysis set population with available data. This information wasn't available for 24 participants.
  Participants
    number analyzed (Participants) | 4083
    Female | 2500
    Male | 1583

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Crohn's Disease Activity Index (CDAI) at Each Visit
Description: The CDAI is a measure of clinical response and remission that was developed for use in clinical trials. The CDAI includes 8 variables encompassing both patient-reported (symptoms, general well-being) and objective (medication usage, laboratory variables, presence of abdominal mass or complications, and weight) variables. For symptoms scores, patients keep track of daily symptoms on a diary card, and the daily symptom scores are summed for the week. Each item in the CDAI is assigned a specific weight, and the weighted values of the items are totaled to produce the CDAI score. Higher CDAI scores indicate greater disease activity; 0 would the lower limit with no set upper limit. The scale for the scores is as follows: < 150 to indicate remission, 150 - 219 to define mildly active disease, 220 - 450 to define moderately active disease, and > 450 to define severely active disease. Negative changes indicate reductions (improvement) in disease activity.
Time Frame: Months 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Effectiveness analyses included all participants with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Crohn's Disease (CD)
Number analyzed (Participants) | 1168
units on a scale
  Month 3 | -117 (117)
  Month 6: number analyzed (Participants) | 992
  Month 6 | -124 (127)
  Month 9: number analyzed (Participants) | 832
  Month 9 | -131 (122)
  Month 12: number analyzed (Participants) | 734
  Month 12 | -137 (125)
  Month 18: number analyzed (Participants) | 620
  Month 18 | -142 (126)
  Month 24: number analyzed (Participants) | 499
  Month 24 | -137 (135)
  Month 30: number analyzed (Participants) | 346
  Month 30 | -145 (119)
  Month 36: number analyzed (Participants) | 259
  Month 36 | -149 (118)
  Month 42: number analyzed (Participants) | 203
  Month 42 | -151 (113)
  Month 48: number analyzed (Participants) | 149
  Month 48 | -153 (109)
  Month 54: number analyzed (Participants) | 108
  Month 54 | -156 (113)
  Month 60: number analyzed (Participants) | 75
  Month 60 | -138 (119)

2. Primary Outcome: Percentage of Full Analysis Set (FAS) Participants in Each CDAI Disease Classification Over Time
Description: The CDAI is a measure of clinical response and remission that was developed for use in clinical trials. The CDAI includes 8 variables encompassing both participant-reported (symptoms, general well-being) and objective (medication usage, laboratory variables, presence of abdominal mass or complications, and weight) variables. For symptoms scores, patients keep track of daily symptoms on a diary card, and the daily symptom scores are summed for the week. Each item in the CDAI is assigned a specific weight, and the weighted values of the items are totaled to produce the CDAI score. Higher CDAI scores indicate greater disease activity; there is no set upper limit. The scale for the scores is as follows: < 150 to indicate remission, 150 - 219 to define mildly active disease, 220 - 450 to define moderately active disease, and > 450 to define severely active disease.
Time Frame: Months 0, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Effectiveness analyses included all participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Crohn's Disease (CD)
Number analyzed (Participants) | 1471
percentage of participants
  Month 0 (Remission) | 12.2
  Month 0 (Mild disease) | 28.8
  Month 0 (Moderate disease) | 54.2
  Month 0 (Severe disease) | 4.8
  Month 3 (Remission): number analyzed (Participants) | 1240
  Month 3 (Remission) | 64.4
  Month 3 (Mild disease): number analyzed (Participants) | 1240
  Month 3 (Mild disease) | 17.4
  Month 3 (Moderate Disease): number analyzed (Participants) | 1240
  Month 3 (Moderate Disease) | 17.2
  Month 3 (Severe Disease): number analyzed (Participants) | 1240
  Month 3 (Severe Disease) | 1.0
  Month 6 (Remission): number analyzed (Participants) | 1066
  Month 6 (Remission) | 67.0
  Month 6 (Mild Disease): number analyzed (Participants) | 1066
  Month 6 (Mild Disease) | 15.3
  Month 6 (Moderate Disease): number analyzed (Participants) | 1066
  Month 6 (Moderate Disease) | 16.6
  Month 6 (Severe Disease): number analyzed (Participants) | 1066
  Month 6 (Severe Disease) | 1.1
  Month 9 (Remission): number analyzed (Participants) | 880
  Month 9 (Remission) | 66.7
  Month 9 (Mild Disease): number analyzed (Participants) | 880
  Month 9 (Mild Disease) | 18.8
  Month 9 (Moderate Disease): number analyzed (Participants) | 880
  Month 9 (Moderate Disease) | 14.2
  Month 9 (Severe Disease): number analyzed (Participants) | 880
  Month 9 (Severe Disease) | 0.3
  Month 12 (Remission): number analyzed (Participants) | 778
  Month 12 (Remission) | 69.8
  Month 12 (Mild Disease): number analyzed (Participants) | 778
  Month 12 (Mild Disease) | 16.2
  Month 12 (Moderate Disease): number analyzed (Participants) | 778
  Month 12 (Moderate Disease) | 13.4
  Month 12 (Severe Disease): number analyzed (Participants) | 778
  Month 12 (Severe Disease) | 0.6
  Month 18 (Remission): number analyzed (Participants) | 665
  Month 18 (Remission) | 72.8
  Month 18 (Mild disease): number analyzed (Participants) | 665
  Month 18 (Mild disease) | 13.2
  Month 18 (Moderate Disease): number analyzed (Participants) | 665
  Month 18 (Moderate Disease) | 13.2
  Month 18 (Severe Disease): number analyzed (Participants) | 665
  Month 18 (Severe Disease) | 0.8
  Month 24 (Remission): number analyzed (Participants) | 536
  Month 24 (Remission) | 70.7
  Month 24 (Mild Disease): number analyzed (Participants) | 536
  Month 24 (Mild Disease) | 14.9
  Month 24 (Moderate Disease): number analyzed (Participants) | 536
  Month 24 (Moderate Disease) | 12.9
  Month 24 (Severe Disease): number analyzed (Participants) | 536
  Month 24 (Severe Disease) | 1.5
  Month 30 (Remission): number analyzed (Participants) | 369
  Month 30 (Remission) | 73.2
  Month 30 (Mild Disease): number analyzed (Participants) | 369
  Month 30 (Mild Disease) | 14.9
  Month 30 (Moderate Disease): number analyzed (Participants) | 369
  Month 30 (Moderate Disease) | 11.7
  Month 30 (Severe Diease): number analyzed (Participants) | 369
  Month 30 (Severe Diease) | 0.3
  Month 36 (Remission): number analyzed (Participants) | 276
  Month 36 (Remission) | 75.4
  Month 36 (Mild Disease): number analyzed (Participants) | 276
  Month 36 (Mild Disease) | 11.2
  Month 36 (Moderate Disease): number analyzed (Participants) | 276
  Month 36 (Moderate Disease) | 13.0
  Month 36 (Severe Disease): number analyzed (Participants) | 276
  Month 36 (Severe Disease) | 0.4
  Month 42 (Remission): number analyzed (Participants) | 220
  Month 42 (Remission) | 74.5
  Month 42 (Mild Disease): number analyzed (Participants) | 220
  Month 42 (Mild Disease) | 12.3
  Month 42 (Moderate Disease): number analyzed (Participants) | 220
  Month 42 (Moderate Disease) | 13.2
  Month 42 (Severe Disease): number analyzed (Participants) | 220
  Month 42 (Severe Disease) | 0.0
  Month 48 (Remission): number analyzed (Participants) | 161
  Month 48 (Remission) | 72.7
  Month 48 (Mild Disease): number analyzed (Participants) | 161
  Month 48 (Mild Disease) | 16.1
  Month 48 (Moderate Disease): number analyzed (Participants) | 161
  Month 48 (Moderate Disease) | 10.6
  Month 48 (Severe Disease): number analyzed (Participants) | 161
  Month 48 (Severe Disease) | 0.6
  Month 54 (Remission): number analyzed (Participants) | 114
  Month 54 (Remission) | 76.3
  Month 54 (Mild Disease): number analyzed (Participants) | 114
  Month 54 (Mild Disease) | 12.3
  Month 54 (Moderate Disease): number analyzed (Participants) | 114
  Month 54 (Moderate Disease) | 11.4
  Month 54 (Severe Disease): number analyzed (Participants) | 114
  Month 54 (Severe Disease) | 0.0
  Month 60 (Remission): number analyzed (Participants) | 79
  Month 60 (Remission) | 68.4
  Month 60 (Mild Disease): number analyzed (Participants) | 79
  Month 60 (Mild Disease) | 15.2
  Month 60 (Moderate Disease): number analyzed (Participants) | 79
  Month 60 (Moderate Disease) | 16.5
  Month 60 (Severe Disease): number analyzed (Participants) | 79
  Month 60 (Severe Disease) | 0.0

3. Primary Outcome: Mean Change From Baseline in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) at Each Visit in FAS Participants
Description: The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) is an abbreviated version of the Inflammatory Bowel Disease (IBD) Questionnaire, a Health-related quality of life (HRQOL) assessment tool for patients with IBD. The SIBDQ utilizes 10 items concerning patient well-being during the last 2 weeks, each of which is scored on a scale of 1 (poor HRQOL) to 7 (optimum HRQOL). The individual sub scores are added to produce the total SIBDQ score. SIBDQ scores range from 10 to 70 with higher values indicating better HRQOL. Positive changes indicate reductions in disease activity.
Time Frame: Months 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Effectiveness analyses included all participants with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Crohn's Disease (CD)
Number analyzed (Participants) | 947
units on a scale
  Month 3 | 10.8 (12.4)
  Month 6: number analyzed (Participants) | 790
  Month 6 | 12.1 (13.2)
  Month 9: number analyzed (Participants) | 658
  Month 9 | 12.6 (13.3)
  Month 12: number analyzed (Participants) | 576
  Month 12 | 13.7 (13.8)
  Month 18: number analyzed (Participants) | 486
  Month 18 | 13.2 (12.9)
  Month 24: number analyzed (Participants) | 373
  Month 24 | 14.7 (14.6)
  Month 30: number analyzed (Participants) | 225
  Month 30 | 14.8 (14.3)
  Month 36: number analyzed (Participants) | 191
  Month 36 | 14.6 (14.8)
  Month 42: number analyzed (Participants) | 161
  Month 42 | 15.4 (13.6)
  Month 48: number analyzed (Participants) | 118
  Month 48 | 16.9 (14.2)
  Month 54: number analyzed (Participants) | 74
  Month 54 | 18.0 (14.4)
  Month 60: number analyzed (Participants) | 70
  Month 60 | 10.2 (13.3)

4. Primary Outcome: Percentage of Participants With Adverse Events (Excluding Serious Adverse Events)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.
  For more details on adverse events please see the AE section below.
Time Frame: Months 0, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Analysis included safety analysis population with incidence of greater than 1% during the study.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Crohn's Disease (CD)
Number analyzed (Participants) | 4107
percentage of participants | 16.7

5. Secondary Outcome: 4.Mean Harvey Bradshaw Index (HBI) in Full Analysis Set (FAS) Participants Over Time
Description: The HBI is a simplified version of the CDAI; HBI scores correlate well with CDAI scores. The HBI consists of 5 items encompassing patient-reported (well-being, symptoms)and objective (presence of abdominal mass or complications) variables. Symptom scores are based on symptom status on the previous day rather than the total of 7 days as for the CDAI. The total HBI score is the sum of the values for each of the five items. Higher HBI scores indicate greater disease activity; 0 would the lower limit with no set upper limit. Scores < 5 indicate remission, 5 - 7 indicate mild disease, 8 - 16 indicate moderate disease, and 16 indicate severe disease. Each HBI unit is equivalent to approximately 27 CDAI units. Higher scores indicate greater disease activity.
Time Frame: Months 0, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Effectiveness analyses included all participants with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Crohn's Disease (CD)
Number analyzed (Participants) | 1621
units on a scale
  Month 0 | 9.3 (4.6)
  Month 3: number analyzed (Participants) | 1481
  Month 3 | 4.8 (4.5)
  Month 6: number analyzed (Participants) | 1296
  Month 6 | 4.5 (4.6)
  Month 9: number analyzed (Participants) | 1097
  Month 9 | 4.2 (4.2)
  Month 12: number analyzed (Participants) | 977
  Month 12 | 4.1 (4.2)
  Month 18: number analyzed (Participants) | 817
  Month 18 | 3.9 (4.1)
  Month 24: number analyzed (Participants) | 696
  Month 24 | 4.1 (4.7)
  Month 30: number analyzed (Participants) | 450
  Month 30 | 3.5 (3.9)
  Month 36: number analyzed (Participants) | 345
  Month 36 | 3.6 (4.0)
  Month 42: number analyzed (Participants) | 265
  Month 42 | 3.9 (3.9)
  Month 48: number analyzed (Participants) | 200
  Month 48 | 3.4 (3.5)
  Month 54: number analyzed (Participants) | 138
  Month 54 | 3.3 (3.6)
  Month 60: number analyzed (Participants) | 103
  Month 60 | 4.0 (3.9)

6. Secondary Outcome: Compliance With the Self-injection Via the Humira®-PEN
Description: Adalimumab will be self-administered by participants using Humira®-PEN. Analysis of compliance was not performed as outlined in the protocol.
Time Frame: Months 0, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Compliance data were not collected.
Arm/Group | Participants With Crohn's Disease (CD)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of study (month 0) through month 60 following the start of treatment with adalimumab.
Description: Analysis included safety analysis population i.e., all participants who received at least 1 dose of adalimumab with evaluable safety data.
Arm/Group | Participants With Crohn's Disease (CD)
Serious Adverse Events (participants affected / at risk) | 548/4107
Other Adverse Events (participants affected / at risk) | 0/4107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Crohn's Disease (CD) (N=4107)
ANAEMIA (Blood and lymphatic system disorders) | 4
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2
CARDIAC ARREST (Cardiac disorders) | 1
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 2
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 1
INNER EAR DISORDER (Ear and labyrinth disorders) | 1
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1
SECONDARY ADRENOCORTICAL INSUFFICIENCY (Endocrine disorders) | 1
GLAUCOMA (Eye disorders) | 1
ULCERATIVE KERATITIS (Eye disorders) | 1
UVEITIS (Eye disorders) | 1
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 5
ABDOMINAL MASS (Gastrointestinal disorders) | 7
ABDOMINAL PAIN (Gastrointestinal disorders) | 17
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 10
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4
ANAL FISSURE (Gastrointestinal disorders) | 1
ANAL FISTULA (Gastrointestinal disorders) | 22
ANAL SKIN TAGS (Gastrointestinal disorders) | 1
ANAL STENOSIS (Gastrointestinal disorders) | 2
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 1
CHRONIC GASTRITIS (Gastrointestinal disorders) | 3
COLONIC FISTULA (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 57
DIARRHOEA (Gastrointestinal disorders) | 7
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1
DUODENAL PERFORATION (Gastrointestinal disorders) | 1
DUODENAL STENOSIS (Gastrointestinal disorders) | 1
ENTEROCOLONIC FISTULA (Gastrointestinal disorders) | 1
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 6
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 4
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1
FLATULENCE (Gastrointestinal disorders) | 1
GASTRIC STENOSIS (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
GASTROINTESTINAL FISTULA (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 3
GASTROINTESTINAL WALL THICKENING (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1
ILEAL STENOSIS (Gastrointestinal disorders) | 25
ILEUS (Gastrointestinal disorders) | 16
ILEUS PARALYTIC (Gastrointestinal disorders) | 2
INGUINAL HERNIA (Gastrointestinal disorders) | 1
INTESTINAL DILATATION (Gastrointestinal disorders) | 4
INTESTINAL FISTULA (Gastrointestinal disorders) | 10
INTESTINAL HAEMATOMA (Gastrointestinal disorders) | 1
INTESTINAL MASS (Gastrointestinal disorders) | 3
INTESTINAL PERFORATION (Gastrointestinal disorders) | 2
INTESTINAL SCARRING (Gastrointestinal disorders) | 1
INTESTINAL STENOSIS (Gastrointestinal disorders) | 34
JEJUNAL STENOSIS (Gastrointestinal disorders) | 1
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 15
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 2
LOCALISED INTRAABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1
MECHANICAL ILEUS (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 7
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 3
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1
PAINFUL DEFAECATION (Gastrointestinal disorders) | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1
RECTAL STENOSIS (Gastrointestinal disorders) | 2
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 3
STOMATITIS (Gastrointestinal disorders) | 1
SUBILEUS (Gastrointestinal disorders) | 17
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1
VOLVULUS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 9
ADVERSE EVENT (General disorders) | 2
CHEST PAIN (General disorders) | 2
CHILLS (General disorders) | 1
EMBOLIA CUTIS MEDICAMENTOSA (General disorders) | 1
FATIGUE (General disorders) | 1
FEELING HOT (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 6
IMPAIRED HEALING (General disorders) | 7
INFLAMMATION (General disorders) | 1
INJECTION SITE HYPERSENSITIVITY (General disorders) | 1
OEDEMA (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
PAIN (General disorders) | 2
PYREXIA (General disorders) | 7
CHOLANGITIS SCLEROSING (Hepatobiliary disorders) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 2
GALLBLADDER PERFORATION (Hepatobiliary disorders) | 1
GALLBLADDER POLYP (Hepatobiliary disorders) | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1
HEPATITIS CHOLESTATIC (Hepatobiliary disorders) | 1
HYDROCHOLECYSTIS (Hepatobiliary disorders) | 1
ALLERGY TO ANIMAL (Immune system disorders) | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 1
ANAPHYLACTIC SHOCK (Immune system disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
SERUM SICKNESS (Immune system disorders) | 1
ABDOMINAL ABSCESS (Infections and infestations) | 5
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1
ABSCESS (Infections and infestations) | 19
ABSCESS INTESTINAL (Infections and infestations) | 7
ABSCESS JAW (Infections and infestations) | 1
ANAL ABSCESS (Infections and infestations) | 24
ANGULAR CHEILITIS (Infections and infestations) | 1
APPENDICITIS PERFORATED (Infections and infestations) | 1
ARTHRITIS BACTERIAL (Infections and infestations) | 1
BARTHOLIN'S ABSCESS (Infections and infestations) | 2
BREAST ABSCESS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 2
CENTRAL NERVOUS SYSTEM VIRAL INFECTION (Infections and infestations) | 1
CHRONIC SINUSITIS (Infections and infestations) | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2
CONJUNCTIVITIS (Infections and infestations) | 1
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 2
DIARRHOEA INFECTIOUS (Infections and infestations) | 1
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 2
ECZEMA INFECTED (Infections and infestations) | 1
ERYSIPELAS (Infections and infestations) | 6
ESCHERICHIA SEPSIS (Infections and infestations) | 1
FOLLICULITIS (Infections and infestations) | 1
FUNGAL INFECTION (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 2
GONORRHOEA (Infections and infestations) | 1
GROIN ABSCESS (Infections and infestations) | 1
HAEMATOMA INFECTION (Infections and infestations) | 1
HELICOBACTER GASTRITIS (Infections and infestations) | 1
HERPES VIRUS INFECTION (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 4
INFECTED FISTULA (Infections and infestations) | 1
INFECTION (Infections and infestations) | 6
INJECTION SITE ABSCESS (Infections and infestations) | 1
LOCALISED INFECTION (Infections and infestations) | 1
LUNG INFECTION (Infections and infestations) | 3
MENINGOCOCCAL SEPSIS (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 4
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1
OPPORTUNISTIC INFECTION (Infections and infestations) | 1
ORAL CANDIDIASIS (Infections and infestations) | 2
OTITIS MEDIA ACUTE (Infections and infestations) | 1
PARONYCHIA (Infections and infestations) | 1
PERIRECTAL ABSCESS (Infections and infestations) | 14
PERITONEAL ABSCESS (Infections and infestations) | 1
PERITONITIS (Infections and infestations) | 1
PERITONITIS BACTERIAL (Infections and infestations) | 1
PERIUMBILICAL ABSCESS (Infections and infestations) | 1
PILONIDAL CYST (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 5
PULMONARY TUBERCULOSIS (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
RECTAL ABSCESS (Infections and infestations) | 6
RENAL ABSCESS (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 2
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1
TONSILLITIS (Infections and infestations) | 1
TONSILLITIS STREPTOCOCCAL (Infections and infestations) | 1
TUBERCULOSIS (Infections and infestations) | 1
TUBO-OVARIAN ABSCESS (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 2
UROSEPSIS (Infections and infestations) | 1
VARICELLA (Infections and infestations) | 1
VULVAL ABSCESS (Infections and infestations) | 1
ABDOMINAL INJURY (Injury, poisoning and procedural complications) | 1
ACCIDENT AT WORK (Injury, poisoning and procedural complications) | 1
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 5
CONCUSSION (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 2
FALL (Injury, poisoning and procedural complications) | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 3
INTESTINAL ANASTOMOSIS COMPLICATION (Injury, poisoning and procedural complications) | 10
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1
PROCEDURAL INTESTINAL PERFORATION (Injury, poisoning and procedural complications) | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1
STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1
STOMAL HERNIA (Injury, poisoning and procedural complications) | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 1
COLONOSCOPY (Investigations) | 4
DIAGNOSTIC PROCEDURE (Investigations) | 2
EMERGENCY CARE EXAMINATION (Investigations) | 1
ENDOSCOPIC RETROGRADE CHOLANGIOPANCREATOGRAPHY (Investigations) | 1
ENDOSCOPY SMALL INTESTINE (Investigations) | 2
ENDOSCOPY UPPER GASTROINTESTINAL TRACT (Investigations) | 1
ENTEROCLYSIS (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
LAPAROSCOPY (Investigations) | 1
NUCLEAR MAGNETIC RESONANCE IMAGING (Investigations) | 1
OESOPHAGOGASTRODUODENOSCOPY (Investigations) | 1
RENAL FUNCTION TEST ABNORMAL (Investigations) | 1
TRANSAMINASES INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 3
CACHEXIA (Metabolism and nutrition disorders) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1
OBESITY (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
ARTHRITIS ENTEROPATHIC (Musculoskeletal and connective tissue disorders) | 2
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
ENTHESOPATHY (Musculoskeletal and connective tissue disorders) | 1
FISTULA (Musculoskeletal and connective tissue disorders) | 10
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
PERIOSTITIS (Musculoskeletal and connective tissue disorders) | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 3
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ANAPLASTIC ASTROCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BURKITT'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLORECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
FOLLICULAR DENDRITIC CELL SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HODGKIN'S DISEASE STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OESOPHAGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PHAEOCHROMOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SEMINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SMALL INTESTINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 1
BASAL GANGLIA INFARCTION (Nervous system disorders) | 1
BRAIN OEDEMA (Nervous system disorders) | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1
CENTRAL NERVOUS SYSTEM INFLAMMATION (Nervous system disorders) | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DYSAESTHESIA (Nervous system disorders) | 1
EPILEPSY (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 3
HEMIPARESIS (Nervous system disorders) | 1
HYPOAESTHESIA (Nervous system disorders) | 1
INTRACRANIAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 2
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
MULTIPLE SCLEROSIS (Nervous system disorders) | 1
SIMPLE PARTIAL SEIZURES (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 2
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
ABORTION (Pregnancy, puerperium and perinatal conditions) | 2
ABORTION EARLY (Pregnancy, puerperium and perinatal conditions) | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 2
DELIVERY (Pregnancy, puerperium and perinatal conditions) | 2
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 8
DEVICE OCCLUSION (Product Issues) | 1
BIPOLAR DISORDER (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 3
SUICIDE ATTEMPT (Psychiatric disorders) | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 1
CALCULUS BLADDER (Renal and urinary disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 2
RENAL COLIC (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
URETERIC STENOSIS (Renal and urinary disorders) | 1
URETEROLITHIASIS (Renal and urinary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
UROGENITAL FISTULA (Renal and urinary disorders) | 1
VESICAL FISTULA (Renal and urinary disorders) | 1
BREAST PAIN (Reproductive system and breast disorders) | 1
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 2
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 10
VAGINAL FISTULA (Reproductive system and breast disorders) | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL TURBINATE HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 1
NEURODERMATITIS (Skin and subcutaneous tissue disorders) | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 3
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 3
RASH (Skin and subcutaneous tissue disorders) | 6
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1
ROSACEA (Skin and subcutaneous tissue disorders) | 1
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1
INADEQUATE DIET (Social circumstances) | 1
ABSCESS DRAINAGE (Surgical and medical procedures) | 19
ADHESIOLYSIS (Surgical and medical procedures) | 1
ANAL FISTULA EXCISION (Surgical and medical procedures) | 6
ANOPLASTY (Surgical and medical procedures) | 1
ANORECTAL OPERATION (Surgical and medical procedures) | 1
APPENDICECTOMY (Surgical and medical procedures) | 1
BLADDER CATHETERISATION (Surgical and medical procedures) | 1
BREAST CONSERVING SURGERY (Surgical and medical procedures) | 1
CAESAREAN SECTION (Surgical and medical procedures) | 1
CANCER SURGERY (Surgical and medical procedures) | 1
CHOLECYSTECTOMY (Surgical and medical procedures) | 4
COLECTOMY (Surgical and medical procedures) | 8
COLECTOMY TOTAL (Surgical and medical procedures) | 1
COLORECTOSTOMY (Surgical and medical procedures) | 1
COLOSTOMY (Surgical and medical procedures) | 1
DEBRIDEMENT (Surgical and medical procedures) | 2
ENTEROSTOMY (Surgical and medical procedures) | 3
FISTULA REPAIR (Surgical and medical procedures) | 14
GALLBLADDER OPERATION (Surgical and medical procedures) | 2
GASTROINTESTINAL DILATION PROCEDURE (Surgical and medical procedures) | 13
HOSPITALISATION (Surgical and medical procedures) | 2
ILEECTOMY (Surgical and medical procedures) | 2
ILEOCOLOSTOMY (Surgical and medical procedures) | 9
ILEOSTOMY (Surgical and medical procedures) | 9
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 1
INTESTINAL ANASTOMOSIS (Surgical and medical procedures) | 7
INTESTINAL FISTULA REPAIR (Surgical and medical procedures) | 5
INTESTINAL OPERATION (Surgical and medical procedures) | 16
INTESTINAL RESECTION (Surgical and medical procedures) | 50
JEJUNECTOMY (Surgical and medical procedures) | 2
JEJUNOSTOMY (Surgical and medical procedures) | 1
LIPOMA EXCISION (Surgical and medical procedures) | 1
MAMMOPLASTY (Surgical and medical procedures) | 1
MASS EXCISION (Surgical and medical procedures) | 2
NASAL SEPTAL OPERATION (Surgical and medical procedures) | 2
OVARIAN CYSTECTOMY (Surgical and medical procedures) | 2
PROCTECTOMY (Surgical and medical procedures) | 1
PROCTOCOLECTOMY (Surgical and medical procedures) | 3
PYLORUS DILATION PROCEDURE (Surgical and medical procedures) | 2
RECTAL FISTULA REPAIR (Surgical and medical procedures) | 2
RESUSCITATION (Surgical and medical procedures) | 1
SHOULDER OPERATION (Surgical and medical procedures) | 1
SIGMOIDECTOMY (Surgical and medical procedures) | 1
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 3
SMALL INTESTINAL RESECTION (Surgical and medical procedures) | 7
STRICTUROPLASTY (Surgical and medical procedures) | 2
SURGERY (Surgical and medical procedures) | 3
THYROID ADENOMA REMOVAL (Surgical and medical procedures) | 1
TOOTH EXTRACTION (Surgical and medical procedures) | 1
TRANSFUSION (Surgical and medical procedures) | 1
TUMOUR EXCISION (Surgical and medical procedures) | 2
TYMPANOPLASTY (Surgical and medical procedures) | 1
URETERIC OPERATION (Surgical and medical procedures) | 1
URINARY TRACT OPERATION (Surgical and medical procedures) | 1
VAGINOPLASTY (Surgical and medical procedures) | 1
WOUND TREATMENT (Surgical and medical procedures) | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 3
DEEP VEIN THROMBOSIS (Vascular disorders) | 2
HYPERTENSION (Vascular disorders) | 2
HYPOTENSION (Vascular disorders) | 1
THROMBOPHLEBITIS (Vascular disorders) | 1
THROMBOSIS (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.